CLINICAL TRIAL: NCT03290430
Title: End Nicotine Dependence (END) Clinic
Brief Title: End Nicotine Dependence Clinic
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3Z17
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
Keywords: Nicotine Dependence; applied behavioral research
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: this is a quasi-experiment, with 4 intervention arms plus options for supplemental intervention support
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group Counseling (Experimental): Participants will be asked to complete a set of surveys that should take about 30 minutes to finish. The surveys will ask questions about the participant, their health history, their desire to quit smoking, and their beliefs and attitudes. There will be 8 sessions over 4 week, each lasting between 1-2 hours. During these sessions, participants will learn about how to quit smoking by changing habits. Sessions may be audio or video taped.
  The study team will use text messaging as a way to keep in contact with all participants. Participants will have the option of getting text-based support throughout the program no matter which session format they chose. Subjects will receive up to 8 weeks of nicotine replacement therapy.
  Interventions: Behavioral: Group Counseling; Behavioral: Texting support; Drug: Nicotine Replacement Therapy
- Individual Counseling (Experimental): Participants will be asked to complete a set of surveys that should take about 30 minutes to finish. The surveys will ask questions about the participant, their health history, their desire to quit smoking, and their beliefs and attitudes. There will be 8 sessions over 4 week, each lasting between 30-45 minutes. During these sessions, participants will learn about how to quit smoking by changing habits. Sessions may be audio or video taped.
  The study team will use text messaging as a way to keep in contact with all participants. Participants will have the option of getting text-based support throughout the program no matter which session format they chose. Subjects will receive up to 8 weeks of nicotine replacement therapy.
  Interventions: Behavioral: Individual Counseling; Behavioral: Texting support; Drug: Nicotine Replacement Therapy
- Telephone Counseling (Experimental): Participants will be asked to complete a set of surveys that should take about 30 minutes to finish. The surveys will ask questions about the participant, their health history, their desire to quit smoking, and their beliefs and attitudes. There will be 8 phone calls over 4 week, each lasting between 30-45 minutes. During these phone calls, participants will learn about how to quit smoking by changing habits. Sessions may be audio taped.
  The study team will use text messaging as a way to keep in contact with all participants. Participants will have the option of getting text-based support throughout the program no matter which session format they chose. Subjects will receive up to 8 weeks of nicotine replacement therapy.
  Interventions: Behavioral: Phone Counseling; Behavioral: Texting support; Drug: Nicotine Replacement Therapy
- Video Counseling (Experimental): Participants will be asked to complete a set of surveys that should take about 30 minutes to finish. The surveys will ask questions about the participant, their health history, their desire to quit smoking, and their beliefs and attitudes. There will be 8 video calls over 4 week, each lasting between 30-45 minutes. During these video calls, participants will learn about how to quit smoking by changing habits. Sessions may be recorded.
  The study team will use text messaging as a way to keep in contact with all participants. Participants will have the option of getting text-based support throughout the program no matter which session format they chose. Subjects will receive up to 8 weeks of nicotine replacement therapy.
  Interventions: Behavioral: Video Counseling; Behavioral: Texting support; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Group Counseling — 8 sessions over 4 weeks. Lasting 1-2 hours each
  Arms: Group Counseling
Behavioral: Individual Counseling — 8 in person sessions over 4 weeks. Lasting 30-45 minutes each
  Arms: Individual Counseling
Behavioral: Phone Counseling — 8 phone sessions over 4 weeks. Lasting 30-45 minutes each
  Arms: Telephone Counseling
Behavioral: Video Counseling — 8 video call sessions over 4 weeks. Lasting 30-45 minutes each
  Arms: Video Counseling
Behavioral: Texting support — Texts with smoking cessation support throughout the program
Drug: Nicotine Replacement Therapy — Participants will receive up to 8 weeks of over-the-counter nicotine replacement therapy
  Other Names: Nicotine Patch; Nicotine Gum; NRT

SUMMARY:
The purpose of this research is to study a smoking cessation program for adult smokers in Northeast Ohio. The study will also look at how different people respond to the program.

DETAILED DESCRIPTION:
Objective 1: To examine the feasibility of conducting an evidence-based, cognitive behavioral therapy (CBT) for tobacco cessation delivered in multiple formats. Participants will have the opportunity to receive a CBT-based tobacco intervention delivered several possible formats (face-to-face, telephone, video-counseling) based on availability and participant preferences. Study participants will be exposed to cognitive-behavioral cessation and relapse prevention strategies, and discuss barriers to cessation, previous quit attempts, risky situations, and benefits observed after quitting. Participants may also complete exercises designed to assist cessation attempts (e.g., mental and behavioral coping skills, cognitive reframing exercise, health benefits of cessation; and no-smoking behavioral contracts). As supplemental treatment, participants may have the option to receive up to 8 weeks of nicotine replacement therapy and text-messaging support.

Objective 2: To examine the rates of smoking abstinence across intervention formats. Investigators will attempt to follow-up with participants for a 6-months after program completion. Investigators will assess point prevalence abstinence for each intervention delivery method.

Objective 3: To assess individual difference variables that influence outcomes. Investigators will examine individual-difference predictors of outcomes, such as readiness to quit, social support, distress, and environmental factors.

ELIGIBILITY:
Inclusion Criteria:

* Current smokers who would like help quitting (≥ 5 cigarettes per day and/or have a breath carbon monoxide (CO) reading of ≥ 8 ppm)
* Able to speak and read English
* Able to engage using at least one of the intervention formats.

Exclusion Criteria:

* Enrollment in another cessation program
* Do not speak and read English
* Do not have access to at least one intervention format
* Have contraindications for NRT
* Do not have contact information (e.g., address, telephone number)
* Are in treatment for substance abuse (e.g., illicit drugs, alcohol abuse)
* They endorse active addiction to another substance (e.g., illicit drugs or alcohol).
* People who self-report having a severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Rate of 24 hour smoking abstinence across intervention | Up to 24 hours after session 1
  Number of participants who did not smoke for 24 hours. Coded as binary (1 = cessation, 0 = smoking)

SECONDARY OUTCOMES:
Rate of 7-day smoking abstinence across intervention | Up to 7 days after session 1
  Number of participants who did not smoke for 7 days (1 = cessation, 0 = smoking)
Rate of 28-day smoking abstinence across intervention | Up to 28 days after session 1
  Number of participants who did not smoke for 28 days (1 = cessation, 0 = smoking)
Average intervention rating | Up to 4 weeks after session 1
  Scaled survey will be used to assess the quality and the content of the intervention [i.e., the extent to which the content was informative, encouraging, attention capturing, credible, applicable to their lives, and comprehensible.]
Sessions completed | Up to 4 weeks after session 1
  Average count of sessions each participant completed (1-8)
Study Retention | Up to 4 weeks after session 1
Nicotine Replacement Therapy (NRT) Completed | Up to 4 weeks after session 1
  Average count of doses of NRT taken by participants

CONTACTS AND LOCATIONS:
Overall Officials: Monica Webb Hooper, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Case Comprehensive Cancer Center, Cleveland, Ohio, United States